CLINICAL TRIAL: NCT00822718
Title: Obestatin Change in Distal Gastrectomy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2004-05-07
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Gastric Cancer Patients Treated by Subtotal Gastrectomy
Keywords: obestatin; ghrelin; stomach cancer; distal gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
According to Seoul cancer registry data (2000), cancer became the leading cause of death in Korea, accounting for 23.9% of all deaths and gastric cancer is the most prevalent malignant neoplasm, comprising 20.8% of all cancers. Korea and some part of Asian countries have the highest incidence of gastric cancer in the world. Therefore, gastrectomy became one of the most common cancer operation in Korea. Thanks to early detection and intervention, the mortality of early gastric cancer drops dramatically and is now believed to be one of the most curable diseases among all the cancers. However, after successful operation and the declaration of cure of the stomach cancer, the patients are left without stomach for all his remaining life. If the patients lose most of his stomach tissue, there are several problems, which include loss of reservoir function for food and indigestion. Besides, loss of appetite is of the paramount importance because the stomach is an important endocrine organ controlling the appetite via gut-brain axis and the main axis is through a hormone called ghrelin, the only orexigenic hormone in human.

Because ghrelin is mainly secreted by the fundus and body, operations such as laryngoscopic Roux-en-Y gastric bypass: (LRYGBP), laryngoscopic-adjustable silicone gastric banding (LASGB) virtually abolish the ghrelin expressing cells. Thus loss of appetite is an inevitable consequence. Then what happens of the plasma ghrelin after Billoth surgery (standard gastric cancer operation) which removes antrum and body of the stomach where ghrelin expressing cells are relatively less distributed? Also puzzling is the fact that after surgery some patients start to gain weight while others continue to lose weight and appetite. Are there ghrelin-expressing cell hyperplasia in the patients who start to gain weight?

The gastrectomy operation which is performed at the investigators institute is Billoth I or II operation. The operation virtually eliminate the half of the body and most of the antrum. If fundus is involved also, proximal gastrectomy is the operation of the choice. Most of the patients who have these operations will lose weight during 1-3 months after surgery, thereafter slowly recover. However, the mechanism of the weight recovery has not been elucidated so far.

To elucidate the mechanism of re-gaining body weight and possible ghrelin expressing cell hyperplasia, the investigators designed the prospective study to investigate the stomach tissue as well as plasma ghrelin in the patients who are going to have Billoth surgery. The items to be investigated include plasma for hormones (ghrelin, leptin, insulin, CCK, PYY), stomach tissue for ghrelin, diet evaluation and body weight (body mass index) changes for 7 months after gastrectomy.

The investigators hope that their study will reveal the valuable information on the body weight recovery and appetite issue. So far the issue of the stomach cancer patients was related to survival issue. However, to lead a comfortable life the quality of life is also very important. The investigators approach will hint the way of surgery which will benefit the patients to live a happy life.

DETAILED DESCRIPTION:
The below is the items to be included in the study.

* diet evaluation: standard three-day diet evaluation table (Dept. of Nutrition)
* body weight and height: BMI .
* ELISA for plasma ghrelin, leptin, insulin, CCK, PYY: whole blood 5 ml in EDTA tube (sampling time: during fasting, around 8 AM-9 AM if possible)
* two biopsy specimen: the same site. Fundus. One for ELISA and one for IHC
* ELISA for tissue ghrelin: frozen in liquid nitrogen
* immunohistochemistry for ghrelin producing cell hyperplasia, Paraffin block cutting for immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

* patients with informed consent
* gastric cancer patients treated by subtotal gastrectomy (without chemotherapy or radiation therapy) : Actually the differentiation of EGC or AGC depend on the depth of invasion. Therefore if the patients are not cachetic because of metastasis or tumor burden, there is no need toe exclude the AGC patients from the study.

Exclusion Criteria:

* patients with chemotherapy or radiation therapy diabetes mellitus: It has been reported that plasma ghrelin is influenced by the insulin. Thus a history of diabetes exclude the enrollment of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine